CLINICAL TRIAL: NCT00997854
Title: Preterm Neonatal Feeding Protocol Comparing Feed Administration Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Sue Ann Smith, MD, Neonatologist, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5376
Record Dates: First submitted 2009-10-15; First posted 2009-10-19 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Feeding Intolerance
Keywords: Feeding; Intolerance; Preterm; Bolus
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 Bolus Feeds (Active Comparator): This group will receive feeds administered by bolus method over no more than 30 minutes per feed.
  Interventions: Other: Length of time for feed administration
- Group 2- Slow Infusion Feeds (Experimental): This group will receive feeds administered by slow infusion over pump for 2 hours.
  Interventions: Other: Length of time for feed administration

INTERVENTIONS:
Other: Length of time for feed administration — Group 1 will consist of babies fed by bolus method, administered over no more than 30 minutes. Group 2 will be fed by slow infusion by pump over 2 hours.

SUMMARY:
Doctors have tried many different methods of feeding to try to decrease feeding intolerance in preterm babies so that they spend less time receiving liquid nutrition and have fewer problems with feeding intolerance.

The purpose of this study is to test two different methods of feeding preterm babies in the hopes of identifying a method that will decrease some of the feeding intolerance that can occur when feeding premature babies.

ELIGIBILITY:
Inclusion Criteria:

* Any infant born at OHSU or transferred in from another facility whose birthweight is greater than 500 grams and less than 1500 grams, and whose gestational age is less than 32 weeks.

Exclusion Criteria:

* Any infant who has major anomalies including but not limited to *gastroschisis

  * omphalocele
  * bowel obstruction or atresia
  * tracheo-esophageal fistula
  * Hirschsprung's Disease
  * congenital diaphragmatic hernia
  * congenital heart disease and other major syndromes
  * infants who have started enteral feeds prior to entering the study
* Any infant whose birth weight is greater than or equal to 1500 grams or less than 500 grams
* Any infant whose gestational age is greater than 32 weeks.

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To compare feeding intolerance between these two groups as defined by the following criteria: the number of times that the signs and symptoms in an infant caused the perception of feeding intolerance with feeds paused for longer than one feeding. | Daily

SECONDARY OUTCOMES:
To compare the number of days it takes the infant to reach full feeds. | After reaching full feeds.
To compare the number of days the infant requires intravenous nutrition. | After reaching full feeds.
To compare the number of days of overall hospitalization duration. | After patient discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Sue Ann Smith, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Sciences University, Portland, Oregon, United States